CLINICAL TRIAL: NCT02072447
Title: A Study to Determine the Absolute Bioavailability of YH4808 Using Simultaneous Oral Therapeutic- and [14C]-Labeled Intravenous Microdoses
Brief Title: Absolute Bioavailability of YH4808 With Accelerator Mass Spectrometry(AMS)-Based Microdose Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Howard Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Microdose_01(YH4808-110(I))
Record Dates: First submitted 2014-02-21; First posted 2014-02-26 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: absolute bioavailability,; microdose,; AMS
MeSH Terms: conditions — Gastroesophageal Reflux

ARMS (1):
- Microdose (Experimental)
  Interventions: Drug: YH4808 PO and [14C]-YH4808 IV

INTERVENTIONS:
Drug: YH4808 PO and [14C]-YH4808 IV

SUMMARY:
This study aims to determine the absolute bioavailability of YH4808 using simultaneous oral therapeutic- and [14C]-labeled intravenous microdoses.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subject aged 20 to 45 at screening
* subjects who have weight over 55 kg with BMI ranged from 20.0 to 25.0
* subjects who decide to participate voluntarily and write a informed consent form

Exclusion Criteria:

* subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* clinically significant allergic disease (except for mild allergic rhinitis)
* subjects who have determined not eligible by screening test (medical history, physical examination, 12-lead ECG, laboratory test, etc) within 28 days of study start
* subjects considered unsuitable for inclusion by the investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (Fpo) | predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 13, 24, 48, 96, 144, 216 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- See also: Webpage of clinical trial center of Seoul National University Hospital — http://ctc.snuh.org